CLINICAL TRIAL: NCT06180824
Title: A Comparative Study of Efficacy and Safety Between Different Dilution of Insulin Infusion in Controlling Blood Sugar Level in ICU Patient
Brief Title: Efficacy and Safety Between Different Dilution of Insulin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mohd Zulfakar Mazlan, MBBS, Associate Prof Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: InsulinUSM
Record Dates: First submitted 2023-12-04; First posted 2023-12-26 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Hyperglycemia
Keywords: insulin; hyperglycemia; diluent; plastic syringe
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- normal saline (No Intervention): Insulin will be diluted with normal saline crystalloid fluid in 50mls syringe and tubing (same product manufacturer). Blood glucose level will be taken from arterial line at presentation or prior to start insulin and checked using glucometer. Then, at 2 hour and 6 hours after initiation of treatment.
- gelafundin (Active Comparator): Insulin will be diluted with gelafundin colloid fluid in 50mls syringe and tubing (same product manufacturer). Blood glucose level will be taken from arterial line at presentation or prior to start insulin and checked using glucometer. Then, at 2 hour and 6 hours after initiation of treatment.
  Interventions: Drug: Gelafundin

INTERVENTIONS:
Drug: Gelafundin — Insulin will be diluted with gelafundin colloid fluid in 50mls syringe and tubing (same product manufacturer).
  Blood glucose level will be taken from arterial line at presentation or prior to start insulin and checked using glucometer. Then, at 2 hour and 6 hours after initiation of treatment.
  Arms: gelafundin

SUMMARY:
Hyperglycemia associated with insulin resistance is common in critically ill patients, even in those nondiabetic patients. Hyperglycaemia or relative insulin deficiency (or both) during critical illness may directly or indirectly confer a predisposition to complications, such as severe infections, polyneuropathy, multiple-organ failure, and death. Tight glycaemic control in adult long-stay critically ill patients using intensive insulin therapy reduces absolute mortality. It has been reported that pronounced hyperglycemia may lead to complications in such patients, although data from controlled trials are lacking. However, target glycaemia may be difficult to achieve in clinical practice. Insulin adsorption onto infusion equipment (e.g., infusion tubing) may affect glucose control, possibly leading to hyperglycemia. In the use of low-level intravenous insulin infusion for treating diabetic hyperglycaemia and ketoacidosis adsorption of insulin to containers or plastic infusion apparatus results in significant losses of 60-80% of insulin in dilute physiological saline solution.

Problem statement & Study rationale

Up to my knowledge, there is no study that demonstrate differences between types of dilution for insulin infusion in ICU patient in Malaysia; thus, this study is aimed to evaluate it. In 2001 it has been reported that intensive insulin therapy (IIT) in surgical intensive care unit (ICU) patients was associated with reduction in mortality and morbidity as well as other associated factors. There is limited study in comparing dilution of insulin in normal saline and other types of diluents.

Other than that, it is important to know which diluent the best is to choose for the management of hyperglycaemia in ICU patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patient admitted to ICU Hospital USM regardless of whether patient intubated or not.
2. Adult patient 18 years old and above.
3. 2 consecutive blood sugar more than 10 mmol/L including patient with diabetic ketoacidosis and hyperosmolar hyperglycaemic state.
4. Within 12 hours from admission.
5. Patient not in high inotropic support and with APACHE II score less than 17.

Exclusion Criteria:

1. Pregnancy.
2. History of any allergic from previous gelafundin infusion or known patient to have allergic towards gelafundin (allergic card, or information from relatives)
3. Post cardiac arrest or prolonged resuscitation.
4. Patient with cardiogenic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood glucose level | At 2 hours
  Mean of blood glucose level
Blood glucose level | At 6 hours
  Mean of blood glucose level

SECONDARY OUTCOMES:
Mortality | 14 days
  Mortality rate
Mortality | 28 days
  Mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Mohd Zulfakar Mazlan, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No